CLINICAL TRIAL: NCT06114225
Title: A Prospective Phase II Clinical Trial on Pre-operative Immunotherapy and Stereotactic Body Radiotherapy Followed by Metastasectomy in Patients With Pulmonary Resectable Recurrence of Osteosarcoma
Brief Title: Pulmonary Resectable Osteosarcoma Treated by Metastasectomy and Pre-operative Immunotherapy and Stereotactic Body Radiotherapy (PROMIS): a Prospective Clinical Trial
Acronym: PROMIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Weibin Zhang, MD, PhD., Chief director of the orthopaedics department, Vice director of the orthpaedic research institute of Shanghai Jiaotong University, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-LLS-221
Record Dates: First submitted 2023-10-03; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Osteosarcoma
Keywords: neoadjuvant immunotherapy; metastasectomy; osteosarcoma; pulmonary metastasis
MeSH Terms: conditions — Osteosarcoma | interventions — Metastasectomy; Gemcitabine; penpulimab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): The participant receive metastasectomy, immunotherapy and Stereotactic Body Radiotherapy (SBRT)
  Interventions: Combination Product: metastasectomy and pre-operative immunotherapy (gemcitabine and penpulimab ) and stereotactic body radiotherapy

INTERVENTIONS:
Combination Product: metastasectomy and pre-operative immunotherapy (gemcitabine and penpulimab ) and stereotactic body radiotherapy — participants first receive concurrent SBRT and penpulimab (PD-1 blockade) and two cycles of GP regimen (gemcitabine d1,d8 and Penpulimab d8 per a 21-day cycle), followed by complete pulmonary metastasectomy. After surgery, participant receive another 4 cycles of GP regimens followed by Penpulimab monotherapy maintenance. The rationale is that pre-operative SBRT could boost the immune microenvironment, leading to a long-term effect of immunotherapy post-metastasectomy and eventually resulting in better long-term survivorship compared to the histological control for pulmonary resectable recurrence of osteosarcoma .

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of pre-operative concurrent Stereotactic Body Radiotherapy (SBRT) and and programmed cell death protein-1 (PD-1) blockade immunotherapy followed by surgical metastasectomy for resectable metastatic osteosarcoma.

DETAILED DESCRIPTION:
Osteosarcoma is a primary bone malignant tumor with strong metastatic potential. About 15%-20% of osteosarcomas are accompanied by lung metastasis when diagnosed, and about 40% of patients develop secondary lung metastasis after radical surgery of the primary lesion. However, pulmonary metastatic osteosarcoma are often insensitive to traditional radiotherapy and chemotherapy. For resectable lung metastases, the preferred treatment is still complete resection of all metastases and the best therapeutic modality and regimens pre- and post-surgical remains unestablished.

With the advent of immunotherapy, many common solid tumors have made substantial progress through immunotherapy after distant metastasis. However, a number of current clinical studies on immunotherapy for osteosarcoma have shown that the effective rate of immunotherapy for osteosarcoma is about 5% to 10% after single agent treatment, making it regarded as one of the "immune cold" tumor, potentially due to the fact that osteosarcoma often lacks immune cell infiltration, and immune cells in tumors are often difficult to be activated or preserve immune memory. However, the investigators have found in our previous clinical observations that a small number of osteosarcoma patients not only have significant effects on immunotherapy, but even have long-term responses. The investigators unexpectedly found that the degree of tumor pro-inflammatory factors and lymphocyte infiltration in the osteosarcoma sample significantly increased after radiotherapy, especially SBRT. The investigators also discovered that the induction of the formation of "tertiary lymphatic structure" within the tumor might be possible through SBRT as a potential sensitization strategy for immunotherapy in osteosarcoma, which is consistent with the recent knowledge of rado-immunotherapy of several solid tumors.

Therefore, the investigators aim to conduct a prospective phase II clinical trial on pre-operative immunotherapy and stereotactic body radiotherapy (SBRT), followed by metastasectomy in patients with pulmonary resectable recurrence of osteosarcoma. To explore the potential mechanisms related to the pre-operative sensitization of immunotherapy, correlative biomarker analysis is to be performed to explore the tumor microenvironment pre- and post- SBRT to pave the way for further precision immunotherapy of bone sarcoma in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed before any trial-related procedures are carried out.
2. Histologically confirmed osteosarcoma, with a diagnosis of pulmonary metastases without the existence of local recurrence (previous re-resection of local recurrence with wide margin is allowed).
3. Resectable pulmonary nodule(s), defined as nodule(s) that are removable by wedge resection/ segmentectomy/lobectomy without necessitating a total pneumonectomy (e.g., nodules immediately adjacent to the main stem bronchus or main pulmonary vessels), and no evidences of malignant pleural effusion.
4. Participants have received at least one standardized systemic treatment regimen at the time of enrollment, and have not received gemcitabine in the past.
5. Patient has adequate pulmonary function eligible for one-staged or two-staged thoracic surgery.
6. Aged no less than 10 years old and no more than 65 years old;
7. For patients ≥16 years old, ECOG score is between 0 and 2 (for patients with amputations, if they can basically take care of themselves and can move freely for more than 50% of their waking hours with the assistance of stretchers, walkers, wheelchairs, etc.) still included);
8. For patients under 16 years old, Lansky score is at least 70 or above (for patients with amputations who are unable to participate in active recreational activities due to amputation, if they can participate in most active recreational activities with the assistance of walkers, wheelchairs, etc., they are still eligible included).
9. The expected survival time is greater than 24 weeks;
10. The majority of the recurrent lesions with an established radiological diagnosis could receive SBRT;
11. Major organ functions meet basic safety standards within 7-14 days before treatment.
12. Women of childbearing age should agree that they must use contraceptive measures (such as intrauterine devices, birth control pills or condoms) during the study and within 6 months after the end of the study; if in doubt, serum or urine tests within 7 days before study enrollment The pregnancy test is negative and the patient must be non-lactating; the male should agree that contraceptive measures must be used during the study period and within 6 months after the end of the study period;
13. If there are recurrent lesions previously treated by surgery, radiofrequency ablation or radiotherapy:

    1. If the image of the metastatic lesion is stable, enrollment is allowed and SBRT is not required for that lesion;
    2. If the metastatic lesion has image progression, if it was previously treated with surgery and SBRT can be performed, enrollment is allowed; if it was previously treated with radiofrequency ablation or radiotherapy, if repeat SBRT can be considered, enrollment is still allowed.

Exclusion Criteria:

1. Diagnosed with malignant diseases other than tumors within 5 years before the first dose;
2. Currently participating in interventional clinical research treatment, or have received other research drugs or used research equipment within 4 weeks before the first dose;
3. Previously received the following therapies: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or drugs targeting another stimulating or synergistic inhibition of T cell receptors (e.g., CTLA-4, OX-40, CD137) drug and secondary resistance to the drug (i.e., the best efficacy evaluation is CR, PR or SD lasting more than 4 months, but secondary tumor resistance develops after treatment).
4. Received systemic systemic treatment with Chinese patent medicines with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, except local use to control pleural effusion) within 2 weeks before the first dose;
5. Active autoimmune disease requiring systemic treatment (such as use of disease-modifying drugs, glucocorticoids, or immunosuppressants) within 2 years before the first dose. Replacement therapies (such as thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency, etc.) are not considered systemic treatments;
6. Are receiving systemic glucocorticoid treatment (excluding nasal spray, inhaled or other route of topical glucocorticoids) or any other form of immunosuppressive therapy within 7 days before the first dose of the study;
7. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
8. Known to be allergic to any components of monoclonal antibody preparations (have experienced grade 3 or above allergic reactions);
9. Have not fully recovered from toxicity and/or complications caused by any intervention before initiating treatment (i.e., ≤Grade 1 or reaching baseline, excluding fatigue or alopecia);
10. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV1/2 antibody positive);
11. Get live vaccine within 30 days before the first dose (cycle 1, day 1);
12. Pregnant or lactating women;
13. Any serious or uncontrollable systemic disease

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
12-month progression-free survival rate (12m-PFSR) | 12 months from recruitment
  The proportion of patients that are progression-free according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), defined as the ratio of patients who have not died or progressed (CR+PR+SD) over the total number of subjects recruited.

SECONDARY OUTCOMES:
Objective response rate (ORR) | From baseline to disease progression, death or the time of metastasectomy, whichever occurs first, up to 3 years after accrual
  Defined as the number of subjects with a best response of (CR+PR)/total number of subjects*100% based on RECISTv1.1 and irRECIST standards respectively
Disease control rate (DCR) | From baseline to disease progression, death or the time of metastasectomy, whichever occurs first, up to 3 years after accrual
  Defined as the number of subjects with a best response of (CR+PR+SD)/total number of subjects*100% based on RECISTv1.1 and irRECIST standards respectively;
Progression-free survival (PFS) | From baseline to disease progression or death, whichever occurs first, up to 3 years after accrual
  Defined as the time from receiving the first study drug to the death or relapse of the subject, assessed by RECISTv1.1 and irRECIST standards respectively, and estimated by the Kaplan-Meier method, including median, quartile and 95% confidence interval
Overall survival (OS) | From baseline until the reported death of the patients due to any causes, up to 3 years after accrual
  defined as the time from receiving the first study drug treatment to the subject's death, estimated by the Kaplan-Meier method, including median, quartile and 95% confidence interval;
Quality of life assessed by patient-reported outcomes (PROs) | From baseline until the reported death of the patients due to any causes, up to 3 years after accrual
  Assessement of the quality of life score using PROs based on EORTC QLQ-C30 scale (adult) or Paediatric Quality of Life Inventory (PedsQL) scale at baseline and at each followed up after treatment.
Number of participants with adverse events | From the first dose of study treatment to 30 days after the last dose of study treatment or before the start day of new anti-cancer drug therapy, whichever occurs first, up to 3 years.
  Number of participants with Treatment emergent adverse events (TEAE) and serious adverse events (SAE). AE was defines as any toxicities in a participant who received study therapy irrespective of the causal relationship. SAE was defined as one of the following: was fatal or life-threatening; resulted in persistent or significant disability/incapacity or inpatient hospitalization or prolongation of existing hospitalization.
The rate of tumor resectability | At the time of metastasectomy, an average of 8~9 weeks
  Tumor resectability is defined as the number of patients undergoing pre-planned metastasectomy divided by the number of patients considered resectable at baseline.
The incidence of peri-operative complications | At the time of metastasectomy, an average of 8~9 weeks
  Peri-operative complications is defined as the incidence of complications during and following metastasectomy surgery

OTHER OUTCOMES:
Exploratory outcome: progression-free survival(PFS) in different subgroups | From baseline to disease progression or death, whichever occurs first, up to 3 years after accrual.
  The PFS for each subgroups in terms of clinicopathological and genomic characteristics (age, gender, histological type, solitary or multiple metastases, unilateral or bilateral metastases, early or late metastases, calcifying or non-calcifying lesions, with or without lesion cavitation, with or without AEs, etc.
Exploratory outcome: the molecular analysis of tumor sample in correlation with the oncological outcome | From baseline to disease progression or death, whichever occurs first, up to 3 years after accrual.
  To explore the molecular correlative relationship between the genomic complexity(i.e. TMB, neoantigen burden, genomic instability) and the therapeutic outcome.
Exploratory outcome: the expression of immune infiltration biomarker of tumor sample in correlation with the oncological outcome. | From baseline to disease progression or death, whichever occurs first, up to 3 years after accrual.
  To explore the tumor microenvironment (immune infiltration, PD-1/PD-L1 expression, immunogenic death, etc.) pre- and post- SBRT, and conduct correlative analysis between these immune microenvironment indexes and the therapeutic outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Weibin Zhang, PhD, MD, Principal Investigator — Ruijin Hospital; Yuhui Shen, PhD, MD, Principal Investigator — Ruijin Hospital; Qiyuan Bao, PhD, MD, Principal Investigator — Ruijin Hospital; Junxiang Wen, PhD, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
individual participant data (IPD) will be available to academic research upon reasonable request, under the local official rules and regulations.